CLINICAL TRIAL: NCT06517979
Title: Development and Prospective Validation of a Digital Pathology-based Artificial Intelligence Diagnostic Model for Pan-cancer Lymphatic Metastasis
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2024-513-01
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Cancer; Lymphatic Metastasis
Keywords: Artificial Intelligence; Lymph Node Metastasis; Digital Pathology; Whole Slide Image
MeSH Terms: conditions — Neoplasms; Lymphatic Metastasis | interventions — Artificial Intelligence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Histopathological slides of formalin-fixed, paraffin-embedded lymph nodes resected from patients with cancer undergoing radical tumor resection and lymph node dissection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with cancer undergoing LND: Patients undergo radical tumor resection and lymph node dissection (LND)
  Interventions: Diagnostic Test: Artificial intelligence (AI)-based diagnostic model

INTERVENTIONS:
Diagnostic Test: Artificial intelligence (AI)-based diagnostic model — Collect pathological slides of resected lymph nodes of the enrolled patients. Digitise these slides into whole-slide images (WSIs). Analyze the WSIs using the AI model to generate diagnostic results (with or without lymphatic metastasis). No intervention to patients would be performed in this diagnostic test study.

SUMMARY:
The goal of this diagnostic test is to develop an artificial intelligence (AI)-based pan-cancer universal diagnostic model for detecting pathological lymph node metastasis (LNM), and prospectively evaluate its apllication value in the real-world clinical practice.

Investigators will compare the diagnostic performance (sensitivity, specificity, etc.) of the AI model and routine pathological report issued by pathologists, to see if the AI model can improve the clinical workflow of pathological evaluation of cancer LNM in in the real world.

DETAILED DESCRIPTION:
Lymph node metastasis (LNM) is a common mode of cancer metastasis, and accurate postoperative pathological lymph node staging is of great significance for further treatment and prognosis assessment. However, the current pathological evaluation of lymph nodes relies on manual examination by pathologists, which has a relatively low diagnostic efficiency and is prone to missed-diagnosis for micro metastatic lesions.

Therefore, investigators are to develope an artificial intelligence (AI)-based diagnostic model for detecting pathological cancer lymph node metastasis based on deep learning algorithms, and evaluate its apllication value in the real-world clinical settings.

This study is a diagnostic test with no intervention measures, planning to collect pathological slides of formalin-fixed, paraffin-embedded lymph nodes resected from the enrolled patients and digitise them into whole-slide images (WSIs). The AI model will analyse the WSIs and generate pixel-level heatmaps and slide-level diagnostic results (with or without LNM). The routine pathological examination will be performed as usual. These two processes will not interfere with each other. And if there are inconsistency in slide-level classification between AI and routine pathological examination, investigators would convene senior pathologists for discussion to make the final decision (immunohistochemistry would be performed if necessary). The final result will be presented to the patient in the form of a pathological report.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cancer, undergoing radical tumor resection and lymph node dissection.
* Patients with complete clinical and pathological information.

Exclusion Criteria:

* The patient refused to participate in this diagnostic test.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with cancer, undergo radical tumor resection and lymph node dissection are planned to be enrolled in this diagnostic test. Histopathological slides of resected pelvic lymph nodes of enrolled patients will be collected and digitised as whole-slide images (WSIs) for the validation of the AI model.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2024-07-26 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
sensitivity | For each enrolled patient, the diagnosis results of AI model will be obtained in servel days after lymph node dissection, and the sensitivity of the AI model will be evaluated through study completion, an average of 3 year.
  the number of correctly diagnosed positive slides (with lymphatic metastasis), to be divided by the number of positive slides in total

SECONDARY OUTCOMES:
specificity | For each enrolled patient, the diagnosis results of AI model will be obtained in servel days after lymph node dissection, and the sensitivity of the AI model will be evaluated through study completion, an average of 3 year.
  the number of correctly diagnosed negative slides (without lymphatic metastasis), to be divided by the number of negative slides in total

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
To protect patient privacy, pathological slide images and other patient-related data are not publicly accessible.